CLINICAL TRIAL: NCT06153771
Title: Description of Changes in NIRS as a Function of Ductus Arteriosus Status in Very Premature Babies Born Before 32 WG at the DIJON University Hospital: Exploratory Prospective, Monocentric, Observational, Descriptive Study
Brief Title: Description of Changes in NIRS as a Function of Ductus Arteriosus Status in Very Premature Babies Born Before 32 WG at the DIJON University Hospital
Acronym: CAPNIRS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: TERNOY-Carriat 2023
Record Dates: First submitted 2023-11-23; First posted 2023-12-01 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Extremely Premature Newborn (Born Before 32 Weeks' Gestation)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Extremely premature newborn: (born before 32 weeks' gestation)
  Interventions: Other: Collection of brain and kidney NIRS measurements; Other: echocardiography

INTERVENTIONS:
Other: Collection of brain and kidney NIRS measurements — (recorded continuously) by a person not involved in the study 30 minutes before echocardiography was performed
Other: echocardiography — on day 2, day 4 and day 7 of life

SUMMARY:
Monitoring patent ductus arteriosus is currently performed using echocardiography, an operator-dependent examination which requires holding the child on their back and which is potentially time-consuming. This test is usually carried out on days 2, 4 and 7 after birth.

NIRS (near-infrared spectroscopy) is a non-invasive method of monitoring tissue oxygen saturation using infrared light.

The aim of the study was to investigate an association between cerebral and renal NIRS data and ductus arteriosus status obtained by echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Parent who has agreed to participate in the study
* Very premature newborn (born before 32 weeks' gestation)
* Hospitalised in the Neonatal Intensive Care Unit at Dijon University Hospital
* Before 48 hours of life

Exclusion Criteria:

* Newborn with congenital heart disease
* Newborn with a congenital renal anomaly
* Newborn with polymalformative syndrome
* Newborn with a skin anomaly
* Newborn with severe circulatory failure unrelated to the ductus arteriosus

Max Age: 48 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Extremely premature newborn (born before 32 weeks' gestation)
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-09-14 (Actual); Study Completion 2024-09-14 (Actual)

PRIMARY OUTCOMES:
The ultrasound status of the ductus arteriosus | On day 2, day 4 and day 7 of life
  (haemodynamically significant open, non-haemodynamically significant open, closed)

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

IPD SHARING:
Plan to Share IPD: No